CLINICAL TRIAL: NCT00708903
Title: A Single Dose, Crossover, Placebo- and Moxifloxacin-Controlled Study of the Effects of HKI-272 on Cardiac Repolarization in Healthy Adult Subjects
Brief Title: Study to Examine the Effect of HKI-272 on Rhythms of the Heart (Cardiac Repolarization)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3144A1-105
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: Thorough QTc study
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): HKI-272
  Interventions: Drug: neratinib
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- 3 (Active Comparator): Moxifloxacin
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: neratinib — HKI-272
  Arms: 1
Other: Placebo — Placebo
  Arms: 2
Drug: Moxifloxacin
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether HKI-272 affects the rhythms of the heart (cardiac repolarization).

ELIGIBILITY:
Inclusion Criteria:

* Men or women of nonchildbearing potential,
* 18-50 years old.
* Healthy as determined by the investigator, including physical examination, laboratory test results, and medical history.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
QTc interval | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (1):
- Tacoma, Washington, United States